CLINICAL TRIAL: NCT04453358
Title: Cystic Fibrosis Remote Monitoring System to Support Resource-Limited Communities
Brief Title: Cystic Fibrosis Remote Monitoring System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Koronis Biomedical Technologies (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R44MD010177 (NIH)
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: This study is a randomized-comparative study investigating the effectiveness of either low-level virtual coaching vs. high-level virtual coaching in improving airway clearance treatment adherence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Interactive coaching (Active Comparator): Airway clearance therapy using goal setting and interactive feedback.
  Interventions: Device: InCourage-Connect
- Standard of care coaching (Active Comparator): Standard of care airway clearance therapy.
  Interventions: Device: InCourage

INTERVENTIONS:
Device: InCourage-Connect — This intervention will provide patients with clearly stated treatment goals and provide them with interactive feedback based on usage date to help support airway clearance therapy adherence.
  Arms: Interactive coaching
Device: InCourage — This intervention will provide standard of care airway clearance therapy with no interactive feedback on treatment goals and usage.
  Arms: Standard of care coaching

SUMMARY:
The objective of this study is to determine if interactive technology (i.e. virtual coaching) that facilitates vest therapy goal setting and provides positive reinforcement will increase adherence to vest therapy for airway clearance in individuals with CF.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a life-limiting multi-system disease primarily characterized by chronic lung infections and pulmonary symptoms such as cough, dyspnea, and chest tightness. Those with CF rely on numerous pharmaceutical and treatment-based therapies as part of their routine care to maintain lung health. Airway clearance, one such treatment-based therapy, uses breathing techniques and various vibrating devices to mobilize lung secretions and is considered a cornerstone of CF care. Vest therapy, a "shaking vest" that applies pressure and high frequency vibrations to the chest wall is the most commonly used technique for airway clearance in the U.S., but adherence to recommended goals for airway clearance is low. Barriers to adherence include the time limitations and unclear goal setting for effective treatment. A previous pilot study by this research team showed that CF patients find the use of airway clearance vests equipped with both pre-set and individually determined programing capabilities as well as electronic monitoring and transmitting capabilities to be acceptable and feasible. Information such as vest-use time, vest pressure measures, programming choices and symptom reporting is captured by these devices and transmitted to health care teams for review as well as provided to patients to provide feedback on treatment goals. This study aims to determine if providing patients with clearly stated treatment goals and the means to monitor and receive positive reinforcing feedback on vest use through interactive technology (i.e. virtual coaching) will improve vest therapy adherence in individuals with CF.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cystic fibrosis
* Be physically capable of and willing to use the study device
* Access to an internet connection
* Access to a mobile device capable of using applications
* Be familiar with how to utilize a mobile device and/or applications
* Self-reported CF-related therapy adherence between 25%-75% on a screening questionnaire

Exclusion Criteria:

* History of solid-organ transplant
* Inability to speak and read the English language
* Any contraindication to vest use for airway clearance

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Airway Clearance Therapy Adherence | 90 days
  Intervention comparison of adherence measurements: a) to prescribed pressure based upon % of time at prescribed pressure and b) to prescribed duration of treatment based upon % of time using the airway clearance device at prescribed duration (weekly capture).

SECONDARY OUTCOMES:
Lung Function | 180 days
  Intervention comparison of pre and post measures of FEV1 and FVC.
Quality of Life Measurement | 180 days
  Intervention comparison based upon pre and post Cystic Fibrosis Questionnaire Revised (CFQ-R).
  Name of categories/domains CFQ-R:
  9 Quality of life domains: Physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions.
  3 symptom scales: Weight, respiratory, and digestion.
  Scaling of items:
  5 distinct 4-point Likert scales (e.g., always/often/ sometime/never)
  Scoring:
  Scores for each domain; after recording, each item is summed to generate a domain score and standardized. Scores range from 0 to 100, with higher scores indicating better health.
CF Respiratory Symptoms | 180 days
  Intervention comparison based upon pre and post CF Respiratory Symptom Score (CRSS) assessment.
  The score evaluates four symptoms: cough, sputum, breathlessness and fatigue. Each symptom is scored from one (mild symptoms) to four (severe symptoms). The total symptom score was the summation of all the four symptoms.
  Scores range from 4 to 16 with 4 being mild to 16 being most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lechtzin, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No